CLINICAL TRIAL: NCT01549873
Title: Anesthesia During Neurophysiologic Monitoring in Scoliosis Patients: Volatile Agents Versus Total Intravenous Anesthesia
Brief Title: Anesthesia During Neurophysiologic Monitoring in Scoliosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Joseph D. Tobias, Chairman, Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB11-00727
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Results first posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Idiopathic Scoliosis
MeSH Terms: interventions — Propofol; Desflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Total intravenous anesthesia (TIVA) (Active Comparator)
  Interventions: Drug: propofol
- Inhaled anesthesia (Active Comparator)
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: propofol — Propofol adjusted to maintain the bispectral index at 40-60.
  Other Names: Diprivan
  Arms: Total intravenous anesthesia (TIVA)
Drug: Desflurane — Desflurane adjusted to maintain the bispectral index at 40-60.
  Other Names: Suprane
  Arms: Inhaled anesthesia

SUMMARY:
When patients have spinal surgery, electrodes are placed on the body to measure motor evoked potentials (MEP) and somatosensory evoked potentials (SSEP). Many hospitals only use IV anesthesia because they feel that measuring MEP and SSEP is easier using IV anesthesia. At this hospital the investigators typically use inhaled anesthesia and are able to successfully measure MEP and SSEP. This is a study to find out if one method of anesthesia is better than the other for measuring MEP and SSEP.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic scoliosis.

Exclusion Criteria:

* Patients with neuromuscular scoliosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph D Tobias, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Total Intravenous Anesthesia (TIVA) | Inhaled Anesthesia
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Total Intravenous Anesthesia (TIVA) | Inhaled Anesthesia | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 13 | 27
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.5 (2.1) | 15.4 (2.4) | 14.9 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Amplitude Required to Elicit the MEP
Description: Compare the data obtained from neuromonitoring including the amplitude required to elicit the MEP from patients receiving general anesthesia with an inhalational anesthetic agent to those receiving total intravenous anesthesia (TIVA).
Time Frame: at time of surgery
Measure: Mean (Standard Deviation); unit: milliamperes
Arm/Group | Total Intravenous Anesthesia (TIVA) | Inhaled Anesthesia
Number analyzed (Participants) | 15 | 14
milliamperes | 307 (72) | 417 (82)

2. Secondary Outcome: Amplitude of the SSEPs
Description: SSEPs (somatosensory evoked potentials) are most commonly elicited by bipolar transcutaneous electrical stimulation applied on the skin over the trajectory of peripheral nerves of the upper limb (e.g., the median nerve) or lower limb (e.g., the posterior tibial nerve), and then recorded from the scalp. The amplitude is the voltage of the electrical stimulation recorded.
Time Frame: day of surgery
Measure: Mean (Standard Deviation); unit: microvolt
Arm/Group | Total Intravenous Anesthesia (TIVA) | Inhaled Anesthesia
Number analyzed (Participants) | 15 | 14
microvolt | 0.83 (0.4) | 0.84 (0.25)

3. Secondary Outcome: Latency of the SSEP's
Description: SSEPs (somatosensory evoked potentials) are most commonly elicited by bipolar transcutaneous electrical stimulation applied on the skin over the trajectory of peripheral nerves of the upper limb (e.g., the median nerve) or lower limb (e.g., the posterior tibial nerve), and then recorded from the scalp. Latency is the time interval between the stimulation and response.
Time Frame: day of surgery
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Total Intravenous Anesthesia (TIVA) | Inhaled Anesthesia
Number analyzed (Participants) | 15 | 14
milliseconds | 27.6 (1.9) | 28.2 (2)

ADVERSE EVENTS:
Arm/Group | Total Intravenous Anesthesia (TIVA) | Inhaled Anesthesia
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes